CLINICAL TRIAL: NCT04423159
Title: Immunogenicity to Cholera Vaccine Within a Population at Risk in Zambia: Mapping the Kinetics of Immune Responses Over Time
Brief Title: Immunological Characteristics of a Population at Risk of Cholera After Oral Cholera Vaccine (CHOVAXIM)
Acronym: CHOVAXIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Infectious Disease Research in Zambia (Other)
Collaborators: Johns Hopkins University (Other); European and Developing Countries Clinical Trials Partnership (EDCTP) (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CHOVAXIM
Record Dates: First submitted 2020-05-26; First posted 2020-06-09 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Diarrhea Infectious
Keywords: Diarrhea; HIV; Vaccines
MeSH Terms: conditions — Dysentery; Diarrhea

STUDY DESIGN:
Intervention Model Description: A pre/post-vaccine study involving a cohort of individuals receiving an oral cholera vaccine in response to a cholera outbreak in the Lukanga Swamps.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- OCV vaccine (Experimental): Shanchol 1.5mL to be administered orally. Each dose contains V.cholerae O1 Inaba El Tor Strain, Inaba classical strain, ogawa classical strain and O139 strain. As well as Thiomersal and a buffer
  Interventions: Biological: OCV Vaccine

INTERVENTIONS:
Biological: OCV Vaccine — 2 doses of OCV were administered to all enrolled participants 1st dose administered at baseline and second dose administered 28 days post 1st dose.

SUMMARY:
The purpose of the study is to find out if individuals who received first and second dose of Oral Cholera Vaccine (OCV) in Lukanga Swamps, Central Province of Zambia have developed protection against future attacks to cholera. The investigators also want to investigate whether vitamin A deficiency and being HIV positive increases the chances of suffering from cholera.

DETAILED DESCRIPTION:
Cholera is caused by toxigenic strains of Vibrio cholerae O1 and O139 and is characterised by sudden onset of acute watery diarrhoea that can lead to severe dehydration and ultimately death if not treated. Zambia, has continued to experience cholera outbreaks in several parts of the country. In order to curb the disease outbreaks, the World Health Organisation (WHO) recommended introducing cholera vaccination as a supplementary cholera control measure together with other prevention and control strategies, in endemic areas as well as in other places at risk for cholera outbreaks. OCV has recently been introduced to Zambia where a large population was vaccinated with 1 dose of Shanchol®, and about 6 months later over 70% individuals traced to receive a second dose.

Considering the annual outbreaks of cholera in Zambia, there is urgent need to determine whether Shanchol® is able to elicit a sufficient and specific immunological response in individuals who received OCV in Zambia. This study will also help the investigator understand whether there are immune response differences based on genetics and may indicate whether some people may need more vaccine regimens than others.

Objective 1: To profile cholera specific antibody status of a population at risk of cholera before and after receiving 1st and 2nd dose of shanchol ® oral cholera vaccine (OCV) Objective 2: To profile and characterize cholera specific B and T lymphocyte phenotypes among the immunized Zambians Objective 3: Develop and evaluate a non-invasive proxy measure of OCV immune responses Objective 4: To measure the protective value of immunizing HIV-infected individuals through measurement of the neutralization capabilities OCV generated antibodies Objective 5: To assess the impact of ABO blood groups on cholera antibody generation

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 18-65 years are eligible to participate.
* Participant is a resident of the study area. Residence was defined as individuals living in the study area for the past 1 year.
* Written consent provided by participant.

Exclusion Criteria:

* Participant aged less than 18 years
* Refuses to consent to participate
* Pregnancy
* Participant has acute medical illness prior to receipt of oral cholera vaccine -Participant has a history of hospitalization for cholera in the past one week

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2016-10-16 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
Vibriocidal | 4 years
  The primary aim of this project is to determine changes in the vibriocidal geometric mean titers at 6, 12, 24, 30, 36, 42 and 48 months (GMT) in participants who receive the second dose of oral cholera vaccine (OCV) at 28 days .

SECONDARY OUTCOMES:
Vibriocidal | 4 years
  Vibriocidal Antibody Response Rates in HIV infected individuals
Vibriocidal | 1 year
  Detection of vibriocidal antibodies in saliva and compare to serum at 1 year post OCV vaccination

CONTACTS AND LOCATIONS:
Locations (1):
- Waya clinic, Kabwe, Central Province, Zambia

IPD SHARING:
Plan to Share IPD: Yes